CLINICAL TRIAL: NCT05587803
Title: Comparison of NeuroSense/NeuroWave and Sedline/Masimo Indices for Measuring Depth of Sedation in the Intensive Care Unit.
Brief Title: Comparison of 2 Depth of Sedation Indices in the Intensive Care Unit
Acronym: PSIWAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22056PSIWAV
Record Dates: First submitted 2022-09-16; First posted 2022-10-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-05

CONDITIONS: RASS-score; Deep Sedation; Post-cardiac Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- study group (Experimental): This arm consists of all the patients that fulfill the inclusion and exclusion-criteria and are therefore suitable for the study. The Neurowave brain monitor is attached on the patients forehead and the study starts. At that moment the included patients are monitored by the Masimo/Sedline en the Neurosense/Neurowave monitor.
  Interventions: Device: Neurowave and Sedline indices in view

INTERVENTIONS:
Device: Neurowave and Sedline indices in view — 3 additional electrodes are attached on the patients forehead. After electrode placement, the indices of both the SEDLINE device and the NEUROWAVE device are noted every 5 seconds for 1 minute

SUMMARY:
In the intensive care unit of the Free University hospital of Brussels, sedated patients are standardly monitored with the Masimo SEDline device to see how deeply a patient is asleep. During this study we want to attach 1 extra device to 30 sedated patients, lying in the intensive care unit. This device, called the NeuroSENSE brain monitor from Neurowave systems, uses a different scale to indicate the ideal depth of sedation. In total, both devices will be hung on a patient for 2 times 35 minutes. At minute 33, a RASS score will be determined in each patient. This score will be determined by talking to the patient or administering a pain stimulus. Based on the reaction of the patient an estimation can be made how deeply a patient is sleeping. Our goal is to find out which device correlates best with the effective clinical state of the patient.

DETAILED DESCRIPTION:
Adequate sedation level is important for patient comfort and safety. As under- and oversedation are common several devices are used that measure the Depth of Anesthesia (DoA). Each device uses its proprietary algorithm to calculate a depth of anesthesia index and each index has its own optimal range. The optimal range for the NeuroSense monitor (NeuroWave Systems inc., Cleveland, OH, USA) is between 40 and 60, while the optimal range for the SEDline monitor (Masimo Corporation; Irvine, CA, USA) is between 25 and 50. When the device indicates a value within these limits, the patient is optimally anesthetized for a surgical procedure. In this study, 30 patients will be monitored simultaneously by both the Neurowave and SedLine devices. The study will determine which device is the most accurate and therefore the most ideal for use in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Sedated patients hospitalized in ICU of the University Hospital of Brussels
* Patients who are monitored with the SEDline/Masimo monitor
* Patients who receive Remifentanil at a maximum concentration of 0,2 μg/kg/min and propofol with a concentration between 0,5-4,0 mg/kg/h
* Age above 18 years

Exclusion Criteria:

* Patients with facial trauma
* Pregnant patients
* Patients who received muscle re-laxants
* Patients in prone position
* Lack of informed consent from the family
* Patients who are hemodynamically unstable
* Patients with neurotrauma or every other neurologic disorder
* Patients post neurosurgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the depth of sedation indices per assigned RASS score using the prediction probability | 33 minutes
  The main objective of the study is to compare the DoA indices of the NeuroSense/NeuroWave monitor and the SEDline/Masimo monitor in sedated patients in ICU. Both values are then correlated with the patient's clinical sedation level by assigning a RASS score to the patient each time. The RASS score stands for Richmond Agitation Sedation Scale and ranges from -5 to +4. A score of -5 stands for a patient who is unresponsive to any stimuli whereas a score of +4 means a highly combative patient. To determine which device correlates best with the clinic, predictive probability will be used. The prediction probability is a value between 0 and 1. A score of 1 corresponds to a correct classification of the DoA in each case. A value of 0 corresponds to a discordance between the clinic and the index value. The device whose predictive probability is closest to 1 correlates best with the clinic and will likely be the best device to use.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Poelaert, MD,PhD, Principal Investigator
Locations (1):
- UZ Brussel, Brussels, Belgium